CLINICAL TRIAL: NCT03896932
Title: Study of Safety and Efficacy of Mini-pool Intravenous Immunoglobulin (MP-IVIG) Prepared by Assiut University Hospital Blood Bank in Primary Immunodeficiency Patients
Brief Title: Minipooled-IVIG in Primary Immunodeficiency Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshaimaa Mokhtar Selim mohamed, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIG in PID
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- minipooled- Intravenous immunoglobulin(MP-IVIG) (Experimental): • MP-IVIG equivalent to 1 g/ kg of standard IVIG over a 6-hour to 8-hour period monthly alternated by standard IVIG for a period of 12 months follow up and the newly diagnosed cases admitted to AUH in the follow up period will be included.
  Interventions: Other: minipooled- Intravenous immunoglobulin(MP-IVIG)

INTERVENTIONS:
Other: minipooled- Intravenous immunoglobulin(MP-IVIG) — The process of MP-IVIG preparation will involve the use of caprylic acid for purification and virus inactivation of Igs from mini-pools of 20 plasma donations collected in our CBTS in AUH. The equipment used for the process comprised disposable blood bags, hemodialyzers, and purification and microbial filters.

SUMMARY:
1. study the pharmacokinetics of mini-pooled intravenous immunoglobulin( MP-IVIG)
2. Study the safety and efficacy of a newly developed preparation of MP-IVIG in children with primary immunodeficiency (PID) :

   * Adverse reaction of MP-IVIG(anaphylaxis and haemolysis)( no or mild or moderate)
   * Prevention of severe bacterial infection
   * Improvement of general health(weight gain and mentality)
   * Integration in to social live
3. Compare the efficacy of MP-IVIG to standard IVIG in children with primary immunodeficiency (PID).

DETAILED DESCRIPTION:
Primary immunodeficiency diseases (PID) are a heterogeneous group of inherited disorders of the immune system, predisposing individuals to recurrent infections, allergy, autoimmunity, and malignancies. Clinical descriptions have already been made for more than 200 PIDs, for which over 150 forms of PID have been molecularly characterized .

A population prevalence of diagnosed PID in the United States at approximately 1 in 1,200 persons.

A part from local registration in some centres there is no national registry of PID in Egypt, and hence, the prevalence of these disorders in the investigator's population is still unknown .

An increasing number of PID are recognized, and effective treatments are possible. Early use of prophylactic antibiotics and replacement immunoglobulin can prevent significant end organ damage and improve long quality of life in these patients .

Immunoglobulin G (IgG) is an essential plasma derived medicine that is lacking in developing countries .IgG shortages leave immune deficient patients without treatment, exposing them to devastating recurrent infections from local pathogens. A simple and practical method for producing IgG from normal plasma collected in developing countries is needed to provide better, faster access to IgG for patients .

Magdy EL-Ekiaby, et al 2010 introduce the concept of small-scale ("minipool") plasma processing methods implementable with minimum infrastructural requirements. They developed viral inactivation and protein purification technologies in single-use equipment to prepare virally safe solvent/detergent-filtered (S/D-F) plasma Producing a 90%pure immunoglobulin fraction in disposable single-use devices for transfusion as well as minipool S/D-F cryoprecipitate to treat bleeding disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age group: children patients under 18 years.
* The study will include patient diagnosed as primary immunodeficiency disease (PID) in Assiut university hospital on standard IVIG therapy.

Exclusion Criteria:

* Patient has SCID.
* Patient with history of severe IVIG side effect.
* Patient with severe immunodeficiency and has severe disseminated infection.
* Patient with renal impairment
* Patient with hepatic cell failure
* Patient with endocrinal abnormalities
* patient with secondary immunodeficiency diseases

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of MP-IVIG assessed by the incidence of acute Serious Bacterial infections(SBIs) | 1 year
  The rate of Acute SBIs for each participant per 1 year will be assessed by questionnaire (Serious Bacterial Infections) include sign and symptoms of acute serious bacterial infections, i.e. bacterial pneumonia, bacteremia/sepsis, bacterial meningitis, osteomyelitis/ septic arthritis, visceral abscess.
Safty of MP-IVIG assessed by percentage of adverse Events | 72 hour after adminstration of MP-IVIG and betwen infusions period
  Overall percentage of adverse events as hemolysis and anaphylaxis headache and other complains that occur during 72 hours of following an infusion of MP-IVIG will be assessed by1) vital sign(pulse,blood pressure,Respiratory rate and temprature 2)Hemolysis by hemoglobin level,LDH,billirubin level.2)lbetwen infusions by home diaries.
Study the pharmacokinetics- MP-IVIG trough levels | predose sample
  MP-IVIG trough level concentration values of serum total IgG pre the MP-IVIG infusion
  (if applicable).
Study the pharmacokinetics MP-IVIG plasma concentration -time curve | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose
  Blood samples for analysis of pharmacokinetics MP-IVIG plasma concentration -time curve were obtained and analysed
Study the pharmacokinetics MP-IVIG half-life | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose
  Blood samples for analysis of pharmacokinetics MP-IVIG haf-life were obtained and analysed
Study the pharmacokinetics MP-IVIG area under the curve | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose
  Blood samples for analysis of pharmacokinetics MP-IVIG haf-life were obtained and analysed
Study the pharmacokinetics MP-IVIG Cmax | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose
  Blood samples for analysis of pharmacokinetics MP-IVIG Cmax were obtained and analysed
Study the pharmacokinetics of MP-IVIG-Tmax. | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose
  Blood samples for analysis of pharmacokinetics MP-IVIG Tmax were obtained and analysed
Study the pharmacokinetics of MP-IVIG elimination rate constant(s). | (1 hour, 2 hours and 1, 2, 3, 7, 14 and 21 days) post-dose
  Blood samples for analysis of pharmacokinetics MP-IVIG elimination rate constant(s) were obtained and analysed

SECONDARY OUTCOMES:
Compare efficacy of MP-IVIG vs standard IVIG by compare incidence of SBIs of both | 1 year
  • Compare the efficacy of MP-IVIG to standard IVIG in children with Primary immunodeficiency disease (PID).

CONTACTS AND LOCATIONS:
Overall Officials: Maha A Mohammed, professor, Study Director — Assiut University
Locations (1):
- Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] El-Ekiaby M, Sayed MA, Caron C, Burnouf S, El-Sharkawy N, Goubran H, Radosevich M, Goudemand J, Blum D, de Melo L, Soulie V, Adam J, Burnouf T. Solvent-detergent filtered (S/D-F) fresh frozen plasma and cryoprecipitate minipools prepared in a newly designed integral disposable processing bag system. Transfus Med. 2010 Feb;20(1):48-61. doi: 10.1111/j.1365-3148.2009.00963.x. Epub 2009 Sep 23. PMID 19778318
- [Background] Boyle JM, Buckley RH. Population prevalence of diagnosed primary immunodeficiency diseases in the United States. J Clin Immunol. 2007 Sep;27(5):497-502. doi: 10.1007/s10875-007-9103-1. Epub 2007 Jun 19. PMID 17577648
- [Background] Reda SM, Afifi HM, Amine MM. Primary immunodeficiency diseases in Egyptian children: a single-center study. J Clin Immunol. 2009 May;29(3):343-51. doi: 10.1007/s10875-008-9260-x. Epub 2008 Nov 11. PMID 19002574
- [Background] Piguet D, Tosi C, Luthi JM, Andresen I, Juge O; Study investigators. Redimune NF Liquid, a ready-to-use, high-concentration intravenous immunoglobulin therapy preparation, is safe and typically well tolerated in the routine clinical management of a broad range of conditions. Clin Exp Immunol. 2008 Apr;152(1):45-9. doi: 10.1111/j.1365-2249.2008.03597.x. Epub 2008 Jan 28. PMID 18241226
- See also: Gathmann B, Grimbacher B, Beauté J, Dudoit Y, Mahlaoui N, Fischer A(2009):. ESID Registry Working Party. The European internet based patient and research database for primary immunodeficiency: results 2006-2008. Clin Exp Immuno. — http://www.ncbi.nlm.nih.gov/pubmed/19630863